CLINICAL TRIAL: NCT03917615
Title: Pelvic Floor Muscle Contraction Among Physiotherapy Students Before and After "Women Health" Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 123/19
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-04

CONDITIONS: Pelvic Floor Muscle Weakness
Keywords: pelvic diaphragm, Physiotherapy students, education

STUDY DESIGN:
Intervention Model Description: 2 groups according to the year of physiotherapy school.
Who Masked: Participant
Masking Description: Participants will not know the aim of study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- after "women health" course (Experimental): The participants will be instructed to contract the pelvic floor muscle
  Interventions: Other: pelvic floor contraction
- before "women health" course (Active Comparator): The participants will be instructed to contract the pelvic floor muscle
  Interventions: Other: pelvic floor contraction

INTERVENTIONS:
Other: pelvic floor contraction — Ultrasound examination will be performed to asses urinary bladder displacement being a marker for pelvic floor muscle function

SUMMARY:
The study aim is to evaluate the ability to correctly contract pelvic floor muscle among physiotherapy students before and after "women health" course. Pelvic floor muscle contraction will be evaluated via transabdominal ultrasound.

DETAILED DESCRIPTION:
Physiotherapy students during their studying in the physiotherapy Bachelor degree program will be examined. Students will be divided into 2 groups according to their year of studying (if they already studied "women health course or not implying 4th year students compared with 1-3 year level students). Each participant will be asked to contract the pelvic floor muscles.

The assessment of pelvic floor contraction will be measured by measuring bladder displacement via abdominal ultrasound. A curved linear array transducer will be placed in the transverse plane immediately suprapubically over the lower abdomen angled at 15-30 degrees from the vertical. Upward movement of the bladder during contraction will be marked as correct contraction. An on screen caliper and measurement tool will be used to measure bladder amount of bladder displacement.

ELIGIBILITY:
Inclusion Criteria:

* healthy students
* willing to participate in the study

Exclusion Criteria:

* has been treated before for pelvic floor rehabilitation
* active urinary tract infection
* pregnancy
* previous abdominal surgeries

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
direction of urinary bladder displacement during contraction | baseline
  upward or downward displacement of urinary bladder will be measured via diagnostic ultrasound
urinary bladder displacement in millimeters | baseline
  bladder displacement will be measured via diagnostic ultrasound using the on screen caliper tool

SECONDARY OUTCOMES:
pelvic floor muscles endurance of contraction in seconds | baseline
  time of muscle contraction will be measured during the last contraction

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PhD, Study Director — University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
the result of the study will be analysed. a paper will be submitted to international journal with study description including methods, examination protocol results
Supporting Information: Study Protocol
Time Frame: one year

REFERENCES:
- [Result] Ben Ami N, Dar G. What is the most effective verbal instruction for correctly contracting the pelvic floor muscles? Neurourol Urodyn. 2018 Nov;37(8):2904-2910. doi: 10.1002/nau.23810. Epub 2018 Aug 28. PMID 30152550